CLINICAL TRIAL: NCT01703637
Title: A Multicenter, Randomized, Double-Blind Comparative Study of Efficacy，Tolerance and Safety Between Sitagliptin ,Vildagliptin and Saxagliptin After 12-week Monotherapy in Drug-naive Adult Patients With Type 2 Diabetes Mellitus
Brief Title: Efficacy and Safety Comparative Study of Sitagliptin,Vildagliptin and Saxagliptin
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Lin Liao (Other)
Responsible Party: Sponsor-Investigator, Lin Liao, chief of endocrinology department at Qianfoshan Hospital, Qianfoshan Hospital
Organization: Qianfoshan Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: qfsnfm-001
Record Dates: First submitted 2012-10-06; First posted 2012-10-10 (Estimated); Last update posted 2016-03-31 (Estimated); Status verified 2016-03

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Sitagliptin; Vildagliptin; Saxagliptin; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Sitagliptin Phosphate; Vildagliptin; saxagliptin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Sitagliptin (Experimental): Drug: sitagliptin sitagliptin 100mg tablet by mouth , once daily for 12 weeks
  Interventions: Drug: Sitagliptin
- Vildagliptin (Experimental): Drug: vildagliptin saxagliptin 50mg tablet by mouth , twice daily for 12 weeks
  Interventions: Drug: Vildagliptin
- Saxagliptin (Experimental): Drug: saxagliptin saxagliptin 5mg tablet by mouth , once daily for 12 weeks
  Interventions: Drug: Saxagliptin

INTERVENTIONS:
Drug: Sitagliptin — * before breakfast：a tablet of sitagliptin; a tablet of vildagliptin's dummy; a tablet of saxagliptin's dummy
  * before dinner：a tablet of sitagliptin's dummy; a tablet of vildagliptin's dummy; a tablet of saxagliptin's dummy
  Other Names: Januvia
  Arms: Sitagliptin
Drug: Vildagliptin — * before breakfast：a tablet of vildagliptin; a tablet of sitagliptin's dummy; a tablet of saxagliptin's dummy
  * before dinner：a tablet of vildagliptin; a tablet of sitagliptin's dummy; a tablet of saxagliptin's dummy
  Other Names: Galvus
  Arms: Vildagliptin
Drug: Saxagliptin — * before breakfast：a tablet of saxagliptin; a tablet of vildagliptin's dummy; a tablet of sitagliptin's dummy
  * before dinner：a tablet of saxagliptin's dummy; a tablet of vildagliptin's dummy; a tablet of sitagliptin's dummy
  Other Names: Onglyza
  Arms: Saxagliptin

SUMMARY:
The purpose of this study is to explore the differences in efficacy and safety of sitagliptin,vildagliptin and saxagliptin and to find which one is more better in treating type 2 diabetes mellitus.

ELIGIBILITY:
Inclusion Criteria:

* signed the informed consent
* diagnosed with T2DM
* women of childbearing potential were required to have a negative urine; pregnancy test,and agreed to use adequate contraception throughout the; study and for up to 4 weeks after completion
* glycosylated hemoglobin ranged in 6.5-9.5%

Exclusion Criteria:

* patients in pregnancy or lactation period
* ever received any kind of oral Hypoglycemic drug in recent 3 months
* patients were currently receiving treatment with a cytochrome P450 3A4 inducer or depressor,a systemic corticosteroid,or a human immunodeficiency virus anti-viral medication
* gastrointestinal surgery that could affect drug absorption
* patients with haemoglobinopathy or rapidly progressing renal disease, or autoimmune skin disorder
* a recent history of alcohol or drug abuse within the past 12 months
* any contraindication listed in the package inserts of the study drugs
* a history of acute or chronic Pancreatitis or currently
* type 1 diabetes; a history of diabetic ketoacidosis or hyperosmolar nonketonic coma
* New York Heart Association class III or IV congestive heart failure; left ventricular ejection fraction ≤ 40%; a major cardiovascular event within the past 6 months
* significant abnormal liver function, defined as aspartate aminotransferase or alanine aminotransferase > 2 times the upper limit of normal or total bilirubin >34 µmol/L (> 2 mg/dL); or a history of positive serologic evidence of infectious liver disease
* clinical signs or symptoms of active liver disease and/or significant abnormal liver function
* patients with any clinically significant abnormality identified on physical examination, electrocardiogram (ECG), or laboratory tests that, in the judgment of the investigator, would compromise the patients' safety or successful participation in the clinical study
* fasting plasma glucose level > 13.3mmol/l
* creatinine clearance rate ≤ 90ml/min

Ages: 18 Years to 78 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2012-10; Primary Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Change From Baseline in Hemoglobin A1c (A1C) Levels at Week 12 | Baseline and Week 12
  Change from baseline reflects the Week 12 value minus the baseline value. A1C represents the percentage of glycosylated hemoglobin

SECONDARY OUTCOMES:
Change From Baseline in Fasting Plasma Glucose (FPG) at Week 12 | Baseline to Week 12
Change From Baseline in 2-hour Postprandial Glucose at Week 12 | Baseline and Week 12
Change From Baseline in Fasting Insulin at Week 12 | Baseline to Week 12
Change From Baseline in Fasting Glucagon at Week 12 | Baseline and Week 12
Change From Baseline in 2-hour Postprandial Insulin at Week 12 | Baseline and Week 12
Change From Baseline in 2-hour Postprandial Glucagon at Week 12 | Baseline and Week 12
Change From Baseline in abdominal perimeter at Week 12 | Baseline and Week 12
Change From Baseline in Body Weight at Week 12 | Baseline and Week 12
Change From Baseline in Fasting Plasma Lipids at Week 12 | Baseline and Week 12
  fasting plasma lipid parameters including total cholesterol(TC), triglyceride(TG) and Low density lipoprotein(LDL)
The Proportion of Patients Achieving A1C < 7% and Achieving A1C<6.5% at Week12 | Baseline and Week 12
The side effect of each drug. | Baseline to week 12

OTHER OUTCOMES:
gene polymorphism study | baseline and week 12
  We will choose 6 mutation types of CYP3A4 common in Chinese,and make blood medicinal concentration assay of participants with these gene types,and then analyse the association between different gene types and the change of glucose level or HbA1c or rate of adverse event.
change from baseline in content of NOS | baseline and week 12

CONTACTS AND LOCATIONS:
Overall Officials: Lin Liao, MD, Study Chair — Qianfoshan Hospital
Locations (8):
- China (8):
  - YuCheng people's hospital, Dezhou, Shandong
  - Hospital of SINOTRUK, Jinan, Shandong
  - Jinan central hospital, Jinan, Shandong
  - The jinan military region general hospital, Jinan, Shandong
  - Qianfoshan Hospital, Jinan, Shandong
  - People's Hospital of Qingdao Chengyang, Qingdao, Shandong
  - Zibo central hospital, Zibo, Shandong
  - Zibo eighth people's hospital, Zibo, Shandong

REFERENCES:
- [Derived] Zhou XJ, Ding L, Liu JX, Su LQ, Dong JJ, Liao L. Efficacy and short-term side effects of sitagliptin, vildagliptin and saxagliptin in Chinese diabetes: a randomized clinical trial. Endocr Connect. 2019 Apr;8(4):318-325. doi: 10.1530/EC-18-0523. PMID 30822272